CLINICAL TRIAL: NCT02559518
Title: Effects of Non-invasive Cerebellar Stimulation on Motor Learning and Cortical Electrical Activity of Healthy Individuals
Brief Title: Non-invasive Cerebellar Stimulation on Motor Learning
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Federal de Pernambuco (Other)
Responsible Party: Principal Investigator, Kátia Monte-Silva, PhD, Universidade Federal de Pernambuco
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: Cerebellum_MotorLearning
Record Dates: First submitted 2015-09-01; First posted 2015-09-24 (Estimated); Last update posted 2018-10-12 (Actual); Status verified 2018-10

CONDITIONS: Healthy
Keywords: Cerebellum; Transcranial Direct Current Stimulation; Repetitive Transcranial Magnetic Stimulation; Motor Learning; Serial Reaction Time Task; HandwritingTask
MeSH Terms: interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (6):
- anodal ctDCS (Experimental): Volunteers will be submitted to non-invasive cerebellar stimulation during serial reaction time task (SRTT).
  Interventions: Device: tDCS; Device: pp-TMS assessment
- cathodal ctDCS (Experimental): Volunteers will be submitted to non-invasive cerebellar stimulation during serial reaction time task (SRTT).
  Interventions: Device: tDCS; Device: pp-TMS assessment
- sham ctDCS (Sham Comparator): Volunteers will be submitted to non-invasive cerebellar stimulation during serial reaction time task (SRTT).
  Interventions: Device: tDCS; Device: pp-TMS assessment
- high frequency c-rTMS (Experimental): Volunteers will be submitted to non-invasive cerebellar stimulation during serial reaction time task (SRTT).
  Interventions: Device: rTMS; Device: pp-TMS assessment
- low frequency c-rTMS (Experimental): Volunteers will be submitted to non-invasive cerebellar stimulation during serial reaction time task (SRTT).
  Interventions: Device: rTMS; Device: pp-TMS assessment
- sham c-rTMS (Sham Comparator): Volunteers will be submitted to non-invasive cerebellar stimulation during serial reaction time task (SRTT).
  Interventions: Device: rTMS; Device: pp-TMS assessment

INTERVENTIONS:
Device: tDCS — Current will be applied by a DC stimulator (NeuroConn Plus, Germany).The active electrode (anode: 5x5 cm²) will be placed over the left cerebellar hemisphere (3 cm lateral to the inion) and the reference (5x7 cm²), over the right arm with current intensity of 2mA, fade in and fade out of 10 seconds, during 20 minutes.
  Arms: anodal ctDCS
Device: tDCS — Current will be applied by a DC stimulator (NeuroConn Plus, Germany). The active electrode (cathode: 5x5 cm²) will be placed over the left cerebellar hemisphere (3 cm lateral to the inion) and the reference (5x7 cm²), over the right arm with current intensity of 2mA, fade in and fade out of 10 seconds, during 20 minutes.
  Arms: cathodal ctDCS
Device: tDCS — Sham ctDCS will be applied using the same electrodes placement and parameter settings of cathodal ctDCS. However, stimulation will last only 30 seconds but volunteers will be with electrodes montage for 20 minutes.
  Arms: sham ctDCS
Device: rTMS — High frequency c-rTMS will be applied through a figure-eight coil connected to a magnetic stimulator (Rapid², Magstim, UK) placed over the left cerebellar hemisphere (3 cm lateral to the inion), tangentially to the scalp and pointing upwards. Protocol: 10Hz, 110% RMT, 33 trains, 50 stimuli per train, intertrain interval of 25 seconds, 1650 stimuli.
  Arms: high frequency c-rTMS
Device: rTMS — Low frequency c-rTMS will be applied through a figure-eight coil connected to a magnetic stimulator (Rapid², Magstim, UK) placed over the left cerebellar hemisphere (3 cm lateral to the inion), tangentially to the scalp and pointing upwards. Protocol: 1Hz, 110% RMT, 1000 stimuli (1 train).
  Arms: low frequency c-rTMS
Device: rTMS — Sham c-rTMS will be performed with low frequency protocol using two coils. The first one - connected to the stimulator (Rapid², Magstim, UK) - will be positioned on a coil support close to the volunteer but not visible. Therefore, characteristic stimulation noises will be audible. The second - disconnected to the stimulator - will be placed over left cerebellar hemisphere.
  Arms: sham c-rTMS
Device: pp-TMS assessment — SICI and ICF will be evaluated through pp-TMS. Subthreshold conditioning stimuli (80% of RMT) and suprathreshold test stimuli (120% of RMT) will be delivered at 2 milliseconds ISI, in order to determine SICI. ICF will be evaluated by MEP average at an ISI of 10 milliseconds. Ten stimuli will be applied at each condition (unconditioned pulse and pairs of stimuli with ISI of 2 and 10 milliseconds). Stimuli order delivery will be pseudo-randomized and SICI and ICF will be expressed as conditioned stimulus percentage regarding an unconditioned stimulus.

SUMMARY:
A crossover trial with healthy volunteers will be conducted. Six sessions will be performed once a week in a counterbalanced order and at least with seven days washout period to minimize carry-over effects. In each session, volunteers will be submitted to: fatigue and attention levels evaluation, cortical brain activity measures through paired pulse transcranial magnetic stimulation (pp-TMS), handwriting test, non-invasive cerebellar stimulation during serial reaction time task (SRTT) and performance perception evaluation.

DETAILED DESCRIPTION:
After given prior informed consent, volunteers will be submitted to six pseudo-randomized sessions using a website (randomization.com) by a non-involved researcher. At study beginning, volunteers will be evaluated through structured questionnaire and baseline SRTT will be performed 24 hours before first session. Each session, will comprise the following experimental sequence:

1. Fatigue and attention levels. It will be measured through an analogue scale graded from 0 to 10, where 0 means lower fatigue or attention levels and 10, the higher fatigue or attention levels.
2. Short intracortical inhibition (SICI) and intracortical facilitation (ICF): it will be evaluated through pp-TMS paradigms (Neurosoft, Russia). Initially, rest motor threshold (RMT) will be determined by finding the lowest stimulator output that elicit motor evoked potential (MEP) around 50 μV (TMS Motor Threshold Assessment Tool -MTAT 2.0 - USA). For RMT measure, a figure-eight coil connected to the magnetic stimulator held manually at 45 degrees from the midline, will be placed over the right primary motor cortex (C4 - 10/20 System). Subthreshold conditioning stimuli (80% of RMT) and suprathreshold test stimuli (120% of RMT) will be delivered at an interstimulus interval (ISI) of 2 milliseconds for SICI and 10 milliseconds for ICF. Ten stimuli will be applied at each condition (unconditioned pulse and pairs of stimuli with ISI of 2 and 10 milliseconds). Stimuli order delivery will be pseudo-randomized and SICI and ICF will be expressed as conditioned stimulus percentage regarding unconditioned stimulus.
3. Handwriting test: volunteers will be instructed to write six words with digital pen using the non-dominant hand on a tablet provided with analysis software system (MovAlyzer, EUA). The task will be performed spontaneously, without any instruction bias during writing activity. Each session has different word sequences but the difficulty level will be maintained (six words, two of them with 4, 6 and 8 letters).
4. Non-invasive cerebellar stimulation + Serial Reaction Time Task: Cerebellar stimulation will be applied during SRTT (online acquisition).

   ctDCS - Electrical current will be delivered through a DC stimulator (NeuroConn Plus, Germany) using a pair of saline-soaked sponge electrodes (surface 25cm² and 35cm²). The active electrode (anode or cathode) will be placed over the left cerebellar area (3 cm lateral to the inion - left cerebellar hemisphere) and the reference, over the right arm with current intensity of 2mA, fade in and fade out of 10 seconds, during 20 minutes. Sham tDCS has been used in several studies to evaluate active tDCS effects. Sham ctDCS will be applied using the same electrodes placement and parameter settings of cathodal ctDCS however, stimulation will last only 30 seconds but volunteers will be with electrodes montage for 20 minutes. Because the device will be automatically turned off without volunteer's perception, early sensations (mild to moderate tingling) on stimulation site will be experienced without inducing any modulatory effects. Moreover, after each ctDCS session, an adverse effects questionnaire will be applied.

   c-rTMS - Initially, the higher cortical representation area (hotspot) of first dorsal interosseous (FDI) muscle will be determined through a figure-eight coil connected to the magnetic stimulator (Rapid², Magstim, UK) held manually and positioned on the scalp (C4 - 10/20 System) at an angle of 45 degrees from the midline pointed to the target muscle (FDI). Thereafter, RMT will be measure. Volunteer will be positioned in front of a computer screen in order to perform SRTT during stimulation. The coil will be placed over left cerebellar hemisphere (3 cm lateral to the inion) tangentially to the scalp and pointing upwards. rTMS protocols was based on previous studies and were adjusted to full-fit safety recommendations and also to be able to realize SRTT simultaneously (online acquisition). Low frequency protocol: 1Hz, 110% RMT, 1000 stimuli (1 train). High frequency protocol: 10Hz, 110% RMT, 33 trains, 50 stimuli per train, intertrain interval of 25 seconds, 1650 stimuli. Sham c-rTMS will be performed with low frequency protocol using two coils. The first one - connected to the stimulator - will be positioned on a coil support close to the volunteer but not visible. Therefore, characteristic stimulation noises will be audible. The second - disconnected to the stimulator - will be placed over left cerebellar hemisphere. After each c-rTMS session, presence of adverse effects will be computed.

   Serial Reaction Time Task (SRTT): it will be performed through software with visual stimuli presented on a computer screen in four different positions. Volunteer must press, with the non-dominant hand, a corresponding key with predetermined fingers as soon as possible when a highlighted star appears on the screen. The test comprises eight blocks with 120 trials each. Implicit motor learning is measured by performance changes between the blocks 5, 6 and 7.
5. Short intracortical inhibition (SICI) and intracortical facilitation (ICF): using the same RTM as before.
6. Handwriting test.
7. Fatigue and attention levels.
8. Performance perception evaluation: in order to correlate stimulation type to the conscious improvement on motor task performance (SRTT and handwriting test) will be asked in the end of each session if the volunteer considers that his motor performance was better, worse or the same as before.

ELIGIBILITY:
Inclusion Criteria:

* Right-handed (assessed by Edinburgh Handedness Inventory)
* Healthy volunteers (self report)
* Absence of neurological and psychiatric diseases
* No history of severe musculoskeletal injury to wrists and fingers
* Without using drugs or neuroactive substances regularly

Exclusion Criteria:

* Pregnancy
* Presence of metallic implant close to the target stimulation area
* Acute eczema under the target stimulation area
* Pacemaker
* History of seizures or epilepsy
* Hemodynamic instability

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2015-09 (Actual); Primary Completion 2016-08 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Changes on implicit motor learning | Six weeks (during stimulation protocol)
  Serial reaction time task will be performed during stimulation protocol and will evaluate implicit motor learning through software with visual stimuli presented on a computer screen in four different positions. Volunteer must press, with the non-dominant hand, a corresponding key with predetermined fingers as soon as possible when a highlighted star appears on the screen. The test comprises eight blocks with 120 trials each.

SECONDARY OUTCOMES:
Changes on cortical brain activity (Intracortical inhibition and facilitation) | Six weeks (before and after stimulation protocol)
  SICI and ICF will be evaluated through pp-TMS. Subthreshold conditioning stimuli (80% of RMT) and suprathreshold test stimuli (120% of RMT) will be delivered at 2 milliseconds ISI, in order to determine SICI. ICF will be evaluated by MEP average at an ISI of 10 milliseconds. Ten stimuli will be applied at each condition (unconditioned pulse and pairs of stimuli with ISI of 2 and 10 milliseconds). Stimuli order delivery will be pseudo-randomized and SICI and ICF will be expressed as conditioned stimulus percentage regarding an unconditioned stimulus.
Changes on explicit motor learning | Six weeks (before and after stimulation protocol)
  Handwriting test is an explicit motor learning measure and will be performed before and after stimulation protocol. Volunteers will be instructed to write six words with digital pen using the non-dominant hand on a tablet provided with analysis software system (MovAlyzer, EUA). The task will be performed spontaneously, without any instruction bias during writing activity.

OTHER OUTCOMES:
Changes on fatigue levels | Six weeks (before and after stimulation protocol)
  It will be measured through an analogue scale graded from 0 to 10, where 0 means lower fatigue levels and 10, the higher fatigue levels.
Changes on performance perception | Six weeks (after each session)
  Performance perception evaluation: in order to correlate stimulation type to the conscious improvement on motor task performance (SRTT and handwriting test) will be asked in the end of each session if the volunteer considers that his motor performance was better, worse or the same as before.
Cerebellar stimulation adverse effects | Six weeks (after each session)
  It will be evaluated through structured questionnaires that include most common stimulation sensations such as headache, tingling, skin redness, etc.
Changes on attention levels | Six weeks (before and after stimulation protocol)
  It will be measured through an analogue scale graded from 0 to 10, where 0 means lower attention levels and 10, the higher attention levels.

CONTACTS AND LOCATIONS:
Overall Officials: Kátia K Monte-Silva, PhD, Study Director — Universidade Federal de Pernambuco
Locations (1):
- Applied Neuroscience Laboratory, Recife, Pernambuco, Brazil